CLINICAL TRIAL: NCT02969733
Title: The Interest of the Xylocaine® and Ketamine on the Per and Postoperative Management of Acute and Chronic Postoperative Pain After Colectomy by Laparoscopy
Brief Title: The Interest of the Xylocaine® and Ketamine on the Management of Acute and Chronic Ain After Colectomy by Laparoscopy
Acronym: KETALIDO
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2009_05/0943; 2009-017682-33 (EudraCT Number)
Record Dates: First submitted 2016-11-14; First posted 2016-11-21 (Estimated); Last update posted 2017-09-12 (Actual); Status verified 2017-09

CONDITIONS: Pain, Postoperative
Keywords: postoperative analgesia; PainMatcher
MeSH Terms: conditions — Pain, Postoperative | interventions — Lidocaine; Ketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Xylocaine (Experimental): intravenous administration
  Interventions: Drug: Xylocaine
- Ketamine (Experimental): intravenous administration
  Interventions: Drug: Ketamine
- isotonic saline serum (Placebo Comparator): isotonic saline serum intravenous administration
  Interventions: Drug: isotonic saline serum intravenous administration

INTERVENTIONS:
Drug: Xylocaine — Xylocaine is administered at a dose of 1.5 mg / kg for induction and then relay by syringe pump at a dose of 1.33 mg / kg / hour will be administered throughout the duration of the intervention and for 24 hours after the end of thereof, to obtain deemed effective plasma concentrations of the order of 0.5 to 5 mcg / mL.
  Arms: Xylocaine
Drug: Ketamine — Ketamine will be administered at a dose of 0.5 mg / kg and then relay by syringe pump at a dose of 0.05 mg / kg / hour for the duration of surgery and 24 hours after the end thereof.
  Arms: Ketamine
Drug: isotonic saline serum intravenous administration
  Arms: isotonic saline serum

SUMMARY:
Recent clinical studies in abdominal surgery have shown that the use of Xylocaine® parenterally intraoperative at plasma concentrations below the toxic threshold of 5 .mu.g / ml, had an analgesic effect and decreased postoperative morphine consumption.

This study aims to evaluate the activity of Xylocaine® and ketamine separately administered parenterally, in terms of postoperative morphine consumption and decrease incidences of postoperative chronic pain at 3 and 6 months after laparoscopic colectomy compared the placebo group.

The evaluation of the intensity of postoperative pain, hyperalgesia perished skin surface scarring) and pain perception threshold by Pain Matcher® confirm or not the predictive nature of these criteria in the occurrence of chronic pain.

ELIGIBILITY:
Inclusion Criteria:

* Surgery: segmental or total colectomy performed by laparoscopy
* Anesthesia state 1 and 3

Exclusion Criteria:

* Patients classified Anesthesia state 4 or 5
* Allergy or intolerance to any of the products used in the protocol
* Creatinine clearance calculated by the Cockcroft formula below 50 ml / min
* Hepatocellular insufficiency
* Severe heart failure
* Peptic ulcer
* Chronic inflammatory bowel disease (IBD)
* Previous history of epilepsy or seizures
* Surgery emergency, palliative surgery, revision surgery
* Chronic pain requiring regular intake of analgesics include opioids
* Patients treated with lidocaine patch
* Psychic Disorder
* Additive Conduct vis-à-vis alcohol or mind-altering substances
* Pregnant or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2011-01; Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Morphine consumption | During the first 24 postoperative hours.

SECONDARY OUTCOMES:
Morphine consumption | All 6 hours during the 48 postoperative hours.
Numeric rating scale score | All 2 hours during the first 24 postoperative hours and all 6 hours during the 48 postoperative hours.
Electric nociception threshold measured by PainMatcher | All 2 hours during the first 24 postoperative hours and all 6 hours during the 48 postoperative hours.
Hyperalgesia of peri-scar (in cm²) with a von Frey filament (pressure of 10 grams | At 2 days after postoperative
Questionnaire Douleur de Saint-Antoine (QDSA) , | at 3 months, at 6 months
  evaluation with validated scores for chronic and neuropathic pains
Questionnaire d'Evaluation des Douleurs Neuropathiques (QEDN), | at 3 months, at 6 months
  evaluation with validated scores for chronic and neuropathic pains
Time physiological function recovery | During the first 24 postoperative hours
  Ability to drink, to eat, to urinate, to walk
Duration of hospital stay | At 5 days after postoperative

CONTACTS AND LOCATIONS:
Overall Officials: Gilles Lebuffe, MD, PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- CHRU, Hôpital Claude Huriez, Lille, France

IPD SHARING:
Plan to Share IPD: No